CLINICAL TRIAL: NCT01885325
Title: Multi-component Intervention to Increase Physical Activity in Preschool Children
Acronym: SHAPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Russell Pate, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00004884; 1R01HD055451 (NIH)
Record Dates: First submitted 2013-05-20; First posted 2013-06-24 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Physical Activity
Keywords: Physical Activity; Sedentary Behavior; Preschool Children
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity Preschool Intervention (Experimental): Preschools randomized to the multi-component physical activity preschool intervention received four major components: Move IN (physical education and other indoor activity programming), Move OUT (recess and structured outdoor activity), Move to Learn (Physical Activity in classroom, academic lessons), and enhancing the social environment to promote Physical Activity.
  Interventions: Other: Physical Activity Preschool Intervention
- Control (No Intervention): The preschools in the control group did not receive the intervention

INTERVENTIONS:
Other: Physical Activity Preschool Intervention — Preschools randomized to the multi-component physical activity preschool intervention received four major components:Move IN (physical education and other indoor activity programming), Move OUT (recess and structured outdoor activity), Move to Learn (Physical activity in classroom, academic lessons), and enhancing the social environment to promote PA.The focus in the physical education classes, recess, daily lessons, and reduction of sedentary time will be on providing activities that 3-to 5-year-old children enjoy.
  Arms: Physical Activity Preschool Intervention

SUMMARY:
The study addresses a critical public health problem, childhood obesity, by testing a physical activity intervention in the types of preschools that millions of children attend. Information gained in this study may lead to adoption of preschool policies and instructional practices that increase physical activity and reduce the risk of obesity in preschool children.

DETAILED DESCRIPTION:
Obesity rates in 3-5 year-old American children have increased dramatically in recent decades. Concurrent with this alarming trend, time spent by young children in preschool settings has increased and their time spent in unstructured play has decreased. Recent studies have shown that children in preschools are engaged primarily in sedentary activities. Nonetheless, few interventions designed to increase PA or decrease sedentary behavior have been evaluated in preschool children. The proposed investigation tested a multicomponent intervention designed to increase physical activity energy expenditure (PAEE) in 3-5 year-old children. Sixteen preschools were randomly assigned to intervention or control groups. 500 children, in two annual waves of ~250 children, participated in the measurement protocol at baseline and after exposure to the intervention for 9 months. Child-level measures included moderate-to-vigorous PA, sedentary behavior, and PAEE measured by accelerometry; height, weight and waist circumference; and demographics. The intervention consisted of four components: Move IN (physical education and other indoor activity programming), Move OUT (recess and structured outdoor activity), Move to Learn (PA in classroom, academic lessons), and enhancing the social environment to promote PA. The study's intervention coordinator worked with the preschool directors, teachers, and assistant teachers to facilitate intervention implementation by providing training, materials, and ongoing support and feedback. An extensive process evaluation documented the extent to which the intervention was implemented. Effects of the intervention on PA, sedentary behavior, PAEE, and weight status were determined. In addition, the study examined factors that associate with change in physical activity, sedentary behavior, physical activity energy expenditure and body mass index during a school year in preschool children.

ELIGIBILITY:
Inclusion Criteria:

* All children from participating K-4 classrooms at the participating schools were invited to participate.

Exclusion Criteria:

* Children were excluded only if they had a condition that would limit data collection using an accelerometer (e.g., non-ambulatory children)

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 708 (Actual)
Dates: Start 2008-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in Minutes of Moderate-to- Vigorous Physical Activity (MVPA) | Measured at baseline and 10 months for each wave of data collection
  MVPA was assessed using an accelerometer. Participants wore the accelerometer during all waking hours for 5 consecutive weekdays. MVPA was determined by applying count cutpoints to the accelerometer data and calculating minutes spent above the MVPA threshold (minutes per hour).

SECONDARY OUTCOMES:
Change in Minutes of Sedentary Behavior | Measured at baseline and 10 months for each wave of data collection
  Sedentary behavior was assessed using an accelerometer. Participants wore the accelerometer during all waking hours for 5 consecutive weekdays. Time spent in sedentary behavior was determined by applying count cutpoints to the accelerometer data and calculating minutes spent below the light activity threshold (minutes per hour).
Change in Physical Activity Energy Expenditure (PAEE) | Measured at baseline and 10 months for each wave of data collection
  PAEE is an expression of the energy expended during physical activity. PAEE was assessed via objective measures of physical activity with accelerometry. Participants wore an accelerometer during all waking hours for 5 consecutive weekdays. PAEE was determined by applying criteria to the accelerometer output and weighting the minutes of activity by MET values appropriate for moderate (4 METs) and vigorous activity (7 METs) in this age group.
Change in Body Mass Index (BMI) | Measured at baseline and 10 months for each wave of data collection
  BMI was calculated from measured height and weight for each child and is reported as kg/m^2. Assessments were made using standard anthropometric procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Russell R Pate, PhD, Principal Investigator — University of South Carolina

REFERENCES:
- [Derived] Pate RR, Brown WH, Pfeiffer KA, Howie EK, Saunders RP, Addy CL, Dowda M. An Intervention to Increase Physical Activity in Children: A Randomized Controlled Trial With 4-Year-Olds in Preschools. Am J Prev Med. 2016 Jul;51(1):12-22. doi: 10.1016/j.amepre.2015.12.003. Epub 2016 Jan 20. PMID 26803357
- [Derived] Pfeiffer KA, Saunders RP, Brown WH, Dowda M, Addy CL, Pate RR. Study of Health and Activity in Preschool Environments (SHAPES): study protocol for a randomized trial evaluating a multi-component physical activity intervention in preschool children. BMC Public Health. 2013 Aug 7;13:728. doi: 10.1186/1471-2458-13-728. PMID 23919808